CLINICAL TRIAL: NCT03840486
Title: Real Time Assessment of Pre-oxygenation Utilizing End-tidal Oxygen Measurements Versus Single Breath End-Tidal Oxygen Measurements in Healthy Volunteers
Brief Title: Pre-oxygenation With Real Time End-tidal Oxygen Measurements Versus Single Breath Measurements
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Steven Lindsey, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00100086
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Rapid Sequence Intubation
Keywords: Emergency department; Intubation; Pre-oxygenation
MeSH Terms: conditions — Emergencies | interventions — Oxygen; Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Non-rebreather mask (NRBM) (Active Comparator): Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor will be placed on the participant's face with the non-rebreather mask (NRBM) overlying the sensor. The participants will be randomized to the order of their treatment sequence as follows: oxygen at 15 liters per minute (LPM) for 3 minutes, at 35 LPM for 3 minutes, or at flush rate (55 LPM) for 3 minutes. The maximal reading at the end of this will be recorded, then the study subjects will be allowed to rest until their EtO2 returns to their baseline. They will then be placed back on NRBM at flush rate, allowed to rise to the maximal reading of the previous step, then do a single breath exhaled EtO2 measurement.
  Interventions: Device: Non-rebreather mask (NRBM); Device: Nasal cannula EtO2 sensor; Drug: Oxygen (NRBM)
- Non-invasive ventilator mask (NIV) (Active Comparator): Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor will be placed on the participant's face with the non-invasive ventilator mask (NIV) overlying the sensor. Participants will be randomized to the order of their treatment sequence as follows: NIV at 40% fraction of inspired oxygen (FiO2) for 3 minutes, NIV at 70% FiO2 for 3 minutes, NIV at 100% FiO2 for 3 minutes, the maximal reading at the end of this trial will be recorded. The study subjects will be allowed to rest until their EtO2 returns to their baseline, then they will be placed back on NIV at 100% FiO2, allowed to rise to the maximal reading of the previous step, then do a single breath exhaled EtO2 measurement.
  Interventions: Device: Non-invasive ventilator mask (NIV); Device: Nasal cannula EtO2 sensor; Drug: Oxygen (NIV)

INTERVENTIONS:
Device: Non-rebreather mask (NRBM) — The non-rebreather mask (NRBM) will be used to assist in the delivery of oxygen. Participants will be placed on NRBM at different flow rates (15 LPM, 35 LPM, or Flush rate at 55 LPM).
  Arms: Non-rebreather mask (NRBM)
Device: Non-invasive ventilator mask (NIV) — The NIV is a non-invasive face (nasal) mask for oxygen delivery. Participants will receive oxygen at 40% FiO2 for 3 minutes, 70% FiO2 for 3 minutes or 100% FiO2 for 3 minutes each.
  Arms: Non-invasive ventilator mask (NIV)
Device: Nasal cannula EtO2 sensor — The nasal cannula EtO2 sensor will be placed on the participant's face under the mask to detect the EtO2 levels.
Drug: Oxygen (NRBM) — Oxygen will be delivered via the NRBM. Participants will receive oxygen at different flow rates (15 LPM, 35 LPM, or flush rate at 55 LPM).
  Arms: Non-rebreather mask (NRBM)
Drug: Oxygen (NIV) — Oxygen will be delivered via the NIV mask. Participants will receive oxygen at 40% FiO2, 70% FiO2 or 100% FiO2 for 3 minutes each.
  Arms: Non-invasive ventilator mask (NIV)

SUMMARY:
This study examines the performance of a nasal cannula end-tidal oxygen (EtO2) measurement as compared to the gold standard of single breath end-tidal oxygen measurements in healthy volunteers. The purpose of this study is to examine the ability of each sensor to predict oxygen levels in real time.

DETAILED DESCRIPTION:
Patients in the Emergency Department (ED) undergoing Rapid Sequence Intubation (RSI) are at risk for serious morbidity and mortality. In order to provide oxygen during the apneic period, it is common practice to provide pre-oxygenation prior to the start of the procedure with high flows of oxygen. Techniques commonly employed to pre-oxygenate ED patients undergoing RSI include high flow oxygen via a non-rebreather mask (NRBM), a self-inflating bag-valve mask (BVM), or non-invasive ventilation (NIV). However, there are currently no studies that explore how to assess the quality of a patient's pre-oxygenation in real time prior to intubation.

Several recent studies that have assessed the use of single breath end-tidal oxygen to assess the effectiveness of various oxygenation strategies. Typically, healthy volunteers are placed on 2 to 3 minutes of a certain pre-oxygenation strategy followed by exhalation of a single breath into an end-tidal oxygen sensor. Higher end-tidal oxygen measurements are used as a marker for pre-oxygenation with higher percentages indicating more complete pre-oxygenation.

A goal EtO2 reading of 90% is typically used to indicate maximal pre-oxygenation. However, this method of assessing pre-oxygenation would be impractical in actual ED patients who are critically ill and may not be able to fully participate in such a measurement. In addition, discontinuing a pre-oxygenation method to obtain a single breath EtO2 reading would be unethical as it would interfere with proper pre-oxygenation in a critically ill patient. A better method would be to examine end-tidal oxygen measurements from patients in real-time as they are being pre-oxygenated. This study will examine the use of a real time nasal cannula EtO2 sensor as compared to the gold standard of a single breath exhalation into a static sensor.

Healthy participants will be randomly assigned to use the non-rebreather mask or the non-invasive ventilator. A baseline EtO2 measurement will be obtained with the nasal cannula EtO2 sensor then the mask the participant was randomized to use will be placed over the nasal cannula EtO2 sensor and oxygenation trials will begin. At the end of each trial a single breath end-tidal oxygen measurement will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and older who are able to consent on their own without a legal representative
* Self-identified as being in good health
* Grossly normal dentition as judged by study investigators
* No self-reported symptoms of upper respiratory infection or other infectious process
* No history of severe pulmonary disease or asthma that requires daily use of an inhaler
* Females participants self-report to not be pregnant at time of study enrollment
* Study subjects will be recruited from within the Department of Emergency Medicine at Grady Memorial Hospital and Emory University Hospital Midtown. Study participants will be drawn from a pool that will include nursing staff, paramedical staff, students, residents, and attending physicians.

Exclusion Criteria:

* Participant does not agree to study enrollment
* Participant cannot tolerate the entire course of non-invasive ventilation required to complete the study
* Participant does not agree to the video recording of the oxygen monitor to ensure proper data transcription

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lindsey, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Grady Memorial Hospital and Emory University Hospital Midtown in Atlanta, Georgia, USA. Participant enrollment began September 24, 2019 and the final study assessment occurred on October 20, 2023.
Groups:
- NIV With Delivery Sequence of NIV at 40% FiO2, NIV at 70% FiO2, and NIV at 100% FiO2: Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor was placed on the participant's face with the non-invasive ventilator mask (NIV) overlying the sensor. Participants were randomized to the order of their treatment sequence to one of six combinations. Participants in this study arm received NIV at 40% fraction of inspired oxygen (FiO2), followed by NIV at 70% FiO2 , and lastly NIV at 100% FiO2. Each trial was 3 minutes and a maximal reading at the end of this trial was recorded. Study participants rested until their EtO2 returned to their baseline, then they were placed back on NIV at 100% FiO2, were allowed to rise to the maximal reading of the previous step, then did a single breath exhaled EtO2 measurement.
  Non-invasive ventilator mask (NIV): The NIV is a non-invasive face (nasal) mask for oxygen delivery.
  Nasal cannula EtO2 sensor: The nasal cannula EtO2 sensor was placed on the participant's face under the mask to detect the EtO2 levels.
  Oxygen (NIV): Oxygen was delivered via the NIV mask. Participants received oxygen at 40% FiO2, 70% FiO2 or 100% FiO2 for 3 minutes each.
- NIV With Delivery Sequence of NIV at 70% FiO2, 40% FiO2, and 100% FiO2: Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor was placed on the participant's face with the non-invasive ventilator mask (NIV) overlying the sensor. Participants were randomized to the order of their treatment sequence to one of six combinations. Participants in this study arm received NIV at 70% fraction of inspired oxygen (FiO2), followed by NIV at 40% FiO2, and lastly NIV at 100% FiO2. Each trial was 3 minutes and a maximal reading at the end of this trial was recorded. Study participants rested until their EtO2 returned to their baseline, then they were placed back on NIV at 100% FiO2, were allowed to rise to the maximal reading of the previous step, then did a single breath exhaled EtO2 measurement.
- NIV With Delivery Sequence of NIV at 100% FiO2, NIV at 70% FiO2, and NIV at 40% FiO2: Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor was placed on the participant's face with the non-invasive ventilator mask (NIV) overlying the sensor. Participants were randomized to the order of their treatment sequence to one of six combinations. Participants in this study arm received NIV at 100% fraction of inspired oxygen (FiO2), followed by NIV at 70% FiO2, and lastly NIV at 40% FiO2. Each trial was 3 minutes and a maximal reading at the end of this trial was recorded. Study participants rested until their EtO2 returned to their baseline, then they were placed back on NIV at 100% FiO2, were allowed to rise to the maximal reading of the previous step, then did a single breath exhaled EtO2 measurement.
- NIV With Delivery Sequence of NIV at 40% FiO2, NIV at 100% FiO2, and NIV at 70% FiO2: Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor was placed on the participant's face with the non-invasive ventilator mask (NIV) overlying the sensor. Participants were randomized to the order of their treatment sequence to one of six combinations. Participants in this study arm received NIV at 40% fraction of inspired oxygen (FiO2), followed by NIV at 100% FiO2, and lastly NIV at 70% FiO2. Each trial was 3 minutes and a maximal reading at the end of this trial was recorded. Study participants rested until their EtO2 returned to their baseline, then they were placed back on NIV at 100% FiO2, were allowed to rise to the maximal reading of the previous step, then did a single breath exhaled EtO2 measurement.
- NIV With Delivery Sequence of NIV at 70% FiO2, NIV at 100% FiO2, and NIV at 40% FiO2: Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor was placed on the participant's face with the non-invasive ventilator mask (NIV) overlying the sensor. Participants were randomized to the order of their treatment sequence to one of six combinations. Participants in this study arm received NIV at 70% fraction of inspired oxygen (FiO2), followed by NIV at 100% FiO2, and lastly NIV at 40% FiO2. Each trial was 3 minutes and a maximal reading at the end of this trial was recorded. Study participants rested until their EtO2 returned to their baseline, then they were placed back on NIV at 100% FiO2, were allowed to rise to the maximal reading of the previous step, then did a single breath exhaled EtO2 measurement.
- NIV With Delivery Sequence of NIV at 100% FiO2, NIV at 40% FiO2, and NIV at 70% FiO2: Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor was placed on the participant's face with the non-invasive ventilator mask (NIV) overlying the sensor. Participants were randomized to the order of their treatment sequence to one of six combinations. Participants in this study arm received NIV at 100% fraction of inspired oxygen (FiO2), followed by NIV at 40% FiO2, and lastly NIV at 70% FiO2. Each trial was 3 minutes and a maximal reading at the end of this trial was recorded. Study participants rested until their EtO2 returned to their baseline, then they were placed back on NIV at 100% FiO2, were allowed to rise to the maximal reading of the previous step, then did a single breath exhaled EtO2 measurement.
- NRBM With Delivery Sequence of Oxygen at 15 LPM, 35 LPM, and 55 LPM: Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor was placed on the participant's face with the non-rebreather mask (NRBM) overlying the sensor. The participants were randomized to the order of their treatment sequence in one of 6 possibilities. Participants in this study arm received oxygen at 15 liters per minute (LPM) for 3 minutes, at 35 LPM for 3 minutes, or at 55 LPM for 3 minutes. All trials were 3 minutes in duration and the maximal reading at the end of each trial was recorded, then the study participants were allowed to rest until their EtO2 returned to their baseline. They were then placed back on NRBM at flush rate (55 LPM), allowed to rise to the maximal reading of the previous step, then do a single breath exhaled EtO2 measurement.
  Non-rebreather mask (NRBM): The non-rebreather mask (NRBM) was used to assist in the delivery of oxygen.
  Nasal cannula EtO2 sensor: The nasal cannula EtO2 sensor was placed on the participant's face under the mask to detect the EtO2 levels.
- NRBM With Delivery Sequence of Oxygen at 15 LPM, 55 LPM, and 35 LPM: Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor was placed on the participant's face with the non-rebreather mask (NRBM) overlying the sensor. The participants were randomized to the order of their treatment sequence in one of 6 possibilities. Participants in this study arm received oxygen at 15 liters per minute (LPM) for 3 minutes, at 55 LPM for 3 minutes, or at 35 LPM for 3 minutes. All trials were 3 minutes in duration and the maximal reading at the end of each trial was recorded, then the study participants were allowed to rest until their EtO2 returned to their baseline. They were then placed back on NRBM at flush rate (55 LPM), allowed to rise to the maximal reading of the previous step, then do a single breath exhaled EtO2 measurement.
- NRBM With Delivery Sequence of Oxygen at 35 LPM, 55 LPM, and 15 LPM: Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor was placed on the participant's face with the non-rebreather mask (NRBM) overlying the sensor. The participants were randomized to the order of their treatment sequence in one of 6 possibilities. Participants in this study arm received oxygen at 35 liters per minute (LPM) for 3 minutes, at 55 LPM for 3 minutes, or at 15 LPM for 3 minutes. All trials were 3 minutes in duration and the maximal reading at the end of each trial was recorded, then the study participants were allowed to rest until their EtO2 returned to their baseline. They were then placed back on NRBM at flush rate (55 LPM), allowed to rise to the maximal reading of the previous step, then do a single breath exhaled EtO2 measurement.
- NRBM With Delivery Sequence of Oxygen at 35 LPM, 15 LPM, and 55 LPM: Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor was placed on the participant's face with the non-rebreather mask (NRBM) overlying the sensor. The participants were randomized to the order of their treatment sequence in one of 6 possibilities. Participants in this study arm received oxygen at 35 liters per minute (LPM) for 3 minutes, at 15 LPM for 3 minutes, or at 55 LPM for 3 minutes. All trials were 3 minutes in duration and the maximal reading at the end of each trial was recorded, then the study participants were allowed to rest until their EtO2 returned to their baseline. They were then placed back on NRBM at flush rate (55 LPM), allowed to rise to the maximal reading of the previous step, then do a single breath exhaled EtO2 measurement.
- NRBM With Delivery Sequence of Oxygen at 55 LPM, 35 LPM, and 15 LPM: Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor was placed on the participant's face with the non-rebreather mask (NRBM) overlying the sensor. The participants were randomized to the order of their treatment sequence in one of 6 possibilities. Participants in this study arm received oxygen at 55 liters per minute (LPM) for 3 minutes, at 35 LPM for 3 minutes, or at 15 LPM for 3 minutes. All trials were 3 minutes in duration and the maximal reading at the end of each trial was recorded, then the study participants were allowed to rest until their EtO2 returned to their baseline. They were then placed back on NRBM at flush rate (55 LPM), allowed to rise to the maximal reading of the previous step, then do a single breath exhaled EtO2 measurement.
- NRBM With Delivery Sequence of Oxygen at 55 LPM, 15 LPM, and 35 LPM: Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor was placed on the participant's face with the non-rebreather mask (NRBM) overlying the sensor. The participants were randomized to the order of their treatment sequence in one of 6 possibilities. Participants in this study arm received oxygen at 55 liters per minute (LPM) for 3 minutes, at 15 LPM for 3 minutes, or at 35 LPM for 3 minutes. All trials were 3 minutes in duration and the maximal reading at the end of each trial was recorded, then the study participants were allowed to rest until their EtO2 returned to their baseline. They were then placed back on NRBM at flush rate (55 LPM), allowed to rise to the maximal reading of the previous step, then do a single breath exhaled EtO2 measurement.
Period: Overall Study
Arm/Group | NIV With Delivery Sequence of NIV at 40% FiO2, NIV at 70% FiO2, and NIV at 100% FiO2 | NIV With Delivery Sequence of NIV at 70% FiO2, 40% FiO2, and 100% FiO2 | NIV With Delivery Sequence of NIV at 100% FiO2, NIV at 70% FiO2, and NIV at 40% FiO2 | NIV With Delivery Sequence of NIV at 40% FiO2, NIV at 100% FiO2, and NIV at 70% FiO2 | NIV With Delivery Sequence of NIV at 70% FiO2, NIV at 100% FiO2, and NIV at 40% FiO2 | NIV With Delivery Sequence of NIV at 100% FiO2, NIV at 40% FiO2, and NIV at 70% FiO2 | NRBM With Delivery Sequence of Oxygen at 15 LPM, 35 LPM, and 55 LPM | NRBM With Delivery Sequence of Oxygen at 15 LPM, 55 LPM, and 35 LPM | NRBM With Delivery Sequence of Oxygen at 35 LPM, 55 LPM, and 15 LPM | NRBM With Delivery Sequence of Oxygen at 35 LPM, 15 LPM, and 55 LPM | NRBM With Delivery Sequence of Oxygen at 55 LPM, 35 LPM, and 15 LPM | NRBM With Delivery Sequence of Oxygen at 55 LPM, 15 LPM, and 35 LPM
Started (Started sequence 1) | 7 | 11 | 10 | 9 | 8 | 8 | 8 | 9 | 8 | 9 | 9 | 9
Completed Sequence 1 | 7 | 10 | 10 | 9 | 8 | 8 | 8 | 9 | 8 | 9 | 9 | 9
Completed Sequence 2 | 7 | 10 | 10 | 9 | 8 | 8 | 8 | 9 | 8 | 9 | 9 | 9
Completed (Completed sequence 3) | 7 | 10 | 10 | 9 | 8 | 8 | 8 | 9 | 8 | 9 | 9 | 9
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes participants who completed the study.
Groups:
- Non-invasive Ventilator Mask (NIV): Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor was placed on the participant's face with the non-invasive ventilator mask (NIV) overlying the sensor. Participants were randomized to the order of their treatment sequence to one of six combinations of NIV at 40% fraction of inspired oxygen (FiO2) for 3 minutes, NIV at 70% FiO2 for 3 minutes, NIV at 100% FiO2 for 3 minutes. The maximal reading at the end of each trial was recorded. The study participants were allowed to rest until their EtO2 returned to their baseline, then they were placed back on NIV at 100% FiO2, allowed to rise to the maximal reading of the previous step, then do a single breath exhaled EtO2 measurement.
- Non-rebreather Mask (NRBM): Prior to the start of the study procedure, a nasal cannula end-tidal oxygen (EtO2) sensor was placed on the participant's face with the non-rebreather mask (NRBM) overlying the sensor. The participants were randomized to the order of their treatment sequence to one of six combinations of oxygen at 15 liters per minute (LPM) for 3 minutes, at 35 LPM for 3 minutes, or at flush rate (55 LPM) for 3 minutes. The maximal reading at the end of each trial was recorded, then the study subjects were allowed to rest until their EtO2 returned to their baseline. They were then placed back on NRBM at flush rate, allowed to rise to the maximal reading of the previous step, then do a single breath exhaled EtO2 measurement.
- Total: Total of all reporting groups
Arm/Group | Non-invasive Ventilator Mask (NIV) | Non-rebreather Mask (NRBM) | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28 [26 to 34] | 27 [25 to 34.5] | 28 [26 to 33.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 37 | 67
  Male | 22 | 15 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 52 | 52 | 104
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 24.7 [23 to 28.2] | 24.9 [21.5 to 28.3] | 24.8 [21.9 to 28.3]
Baseline Single Breath End Tidal Oxygen (EtO2%) [Median (Inter-Quartile Range); unit: percent of oxygenation] | 16.8 [16.1 to 17.3] | 16.8 [16.0 to 17.8] | 16.8 [16.1 to 17.5]

OUTCOME MEASURES:

1. Primary Outcome: Real Time and Single Breath End-tidal (EtO2) Measurements
Description: Real-time end-tidal oxygen measurements as measured with a nasal cannula (NC) and single-breath (SB) end-tidal oxygen measurements across increasing oxygen concentrations and flow rates for the non-invasive ventilation (NIV) and non-rebreather mask (NRBM) study arms.
Time Frame: After each 3 minute treatment level
Population: This analysis includes participants who completed all three intervention levels.
Measure: Median (Inter-Quartile Range); unit: percentage of end-tidal oxygen
Groups:
- NIV at 40% FiO2: Participants receiving non-invasive ventilator mask (NIV) at 40% fraction of inspired oxygen (FiO2) for 3 minutes.
- NIV at 70% FiO2: Participants receiving non-invasive ventilator mask (NIV) at 70% fraction of inspired oxygen (FiO2) for 3 minutes.
- NIV at 100% FiO2: Participants receiving non-invasive ventilator mask (NIV) at 100% fraction of inspired oxygen (FiO2) for 3 minutes.
- NRBM at 15 LPM: Participants receiving non-rebreather Mask (NRBM) at 15 liters per minute (LPM) for 3 minutes.
- NRBM at 35 LPM: Participants receiving non-rebreather Mask (NRBM) at 35 liters per minute (LPM) for 3 minutes.
- NRBM at 55 LPM: Participants receiving non-rebreather Mask (NRBM) at 55 liters per minute (LPM) for 3 minutes.
Arm/Group | NIV at 40% FiO2 | NIV at 70% FiO2 | NIV at 100% FiO2 | NRBM at 15 LPM | NRBM at 35 LPM | NRBM at 55 LPM
Number analyzed (Participants) | 52 | 52 | 52 | 52 | 52 | 52
percentage of end-tidal oxygen
  Nasal cannula end-tidal oxygen measurement | 34 [33 to 35.8] | 63 [61 to 64] | 92 [91 to 93] | 58.5 [48.3 to 66] | 79 [72.3 to 84.8] | 87.5 [83 to 91]
  Single-breath end-tidal oxygen measurement | 33.1 [29.9 to 34.6] | 58.4 [52.2 to 61.5] | 84.6 [73.7 to 88.1] | 44.9 [38.7 to 50.1] | 60.8 [51.4 to 69.4] | 70.5 [60.3 to 82.1]

2. Secondary Outcome: Time to Maximum End-tidal Oxygen (EtO2) Nasal Cannula Measurement (TmaxNC)
Description: Time required to reach 3-minute nasal cannula end-tidal oxygen (EtO2) reading for the single-breath (SB) EtO2 measurement at TmaxNC for the non-invasive ventilation (NIV) and non-rebreather mask (NRBM) arms.
Time Frame: Up to 3 minutes
Population: This analysis includes participants who completed all three intervention levels.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Non-invasive Ventilator Mask (NIV) | Non-rebreather Mask (NRBM)
Number analyzed (Participants) | 52 | 52
seconds | 126 [107.2 to 144.8] | 100 [88.5 to 111.5]

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time of the intervention and continuing through the end of the intervention, on Day 1 of the study.
Groups:
- NIV at 40% FiO2: Participants receiving non-invasive ventilator mask (NIV) at 40% FiO2
- NIV at 70% FiO2: Participants receiving NIV at 70% FiO2
- NIV at 100% FiO2: Participants receiving NIV at 100% FiO2
- NRBM at 15 LPM: Participants receiving non-rebreather Mask (NRBM) at 15 liters per minute (LPM)
- NRBM at 35 LPM: Participants receiving NRBM at 35 LPM
- NRBM at 55 LPM: Participants receiving NRBM at 55 LPM
Arm/Group | NIV at 40% FiO2 | NIV at 70% FiO2 | NIV at 100% FiO2 | NRBM at 15 LPM | NRBM at 35 LPM | NRBM at 55 LPM
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53 | 0/52 | 0/52 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/53 | 0/52 | 0/52 | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/53 | 0/52 | 0/52 | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT03840486/Prot_SAP_001.pdf